CLINICAL TRIAL: NCT02279316
Title: Home Exercise, Vitamin D and Dalcroze Eurhythmics for Seniors With Mild Cognitive Impairment (MCI) or Mild Dementia
Brief Title: Move for Your Mind - Pilot Trial
Acronym: MFYM - P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Waid City Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SNCTP000000580
Record Dates: First submitted 2014-10-04; First posted 2014-10-31 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Mild Cognitive Impairment; Mild Dementia; Fall Prevention
Keywords: Dalcroze eurhythmics; home exercise; vitamin D; mild cognitive impairment; MCI; mild dementia
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Jaques-Dalcroze eurhythmics (Experimental): Jaques-Dalcroze eurhythmics (60min/wk) + 800 IU Vitamin D3
  Interventions: Drug: Vi-De 3; Other: Jaques-Dalcroze eurhythmics
- Home exercise program (Experimental): Home exercise strength program (3x30min/wk) + 800 IU vitamin D
  Interventions: Drug: Vi-De 3; Other: Home exercise program
- Vitamin D only (Other): 800 IU Vi-De 3
  Interventions: Drug: Vi-De 3

INTERVENTIONS:
Drug: Vi-De 3 — All participants receive a dose of 800 IU vitamin D3 per day as a standard of care. 800 IU Vitamin D is the dose that is currently recommended by the Swiss Health Department (Bundesamt für Gesundheit) for seniors over 60.
  Other Names: Vitamin D, cholecalciferol
Other: Jaques-Dalcroze eurhythmics — The Jaques-Dalcroze eurhythmics method includes different courses of motion (multi-task exercises) that are conducted to the rhythm of improvised piano music. A session starts with a short warm-up that includes simple exercises to get body and mind prepared for the rest of the exercise session. The complexity of the exercises increases gradually during the session: starting with single tasks and then combining them into a multi-task exercise gradually increasing complexity.
  Arms: Jaques-Dalcroze eurhythmics
Other: Home exercise program — The home exercise program is a strengthening program that will consist of five simple exercises.
  Arms: Home exercise program

SUMMARY:
Move for your mind is a single blind, 3-arm randomized controlled clinical pilot trial. The study aims to test the effect of a weekly Dalcroze eurhythmics program (arm 1) and a home strength exercise program (arm 2) against control (no exercise) on the rate of falling, quality of life, gait performance and cognitive function. All groups receive vitamin D. In addition the study shall test the feasibility of the recruitment and the interventions in this target population.

The study includes 60 seniors, age 65 and older, with mild cognitive impairment or mild dementia. Participants are recruited by the memory clinic of City Hospital Waid.

During the 12 months follow-up, participants will have 3 clinical visits (baseline, 6 and 12 month). Despite major efforts the target population is very difficult to recruit and adherence to treatment is low. We therefore decided to stop recruitment and to use this trial as a pilot trial for future clinical trials of the same topic.

DETAILED DESCRIPTION:
Primary objective To test whether the Jaques-Dalcroze eurhythmics program (1 hour a week for 12 months) and/or the simple home exercise program (3 × 30 min a week for 12 months) will decrease rate of falls in seniors with MCI or mild dementia compared with the control group.

Secondary objectives Objective 1: To test whether the Jaques-Dalcroze eurhythmics program (1 hour a week for 12 months) and/or the simple home exercise program (3 × 30 min a week for 12 months) decreases 12-month risk of falling at least once in seniors with MCI or mild dementia compared with the control group.

Objective 2: To test whether the Jaques-Dalcroze eurhythmics program (1 hour a week for 12 months) and/or the simple home exercise program (3 × 30 min a week for 12 months) improves cognitive func-tion and alertness in seniors with MCI or mild dementia compared with the control group.

Objective 3: To test whether the Jaques-Dalcroze eurhythmics program (1 hour a week for 12 months) and/or the simple home exercise program (3 × 30 min a week for 12 months) decreases gait variability in seniors with MCI or mild dementia compared with the control group.

Objective 4: To test whether the Jaques-Dalcroze eurhythmics program (1 hour a week for 12 months) and/or the simple home exercise program (3 × 30 min a week for 12 months) improves quality of life in seniors with MCI or mild dementia compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 65+ years
* Diagnosed with MCI or mild dementia by the memory clinic of City Hospital Waid

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rate of falls (any falls, low trauma falls, injurious falls) during 12 month follow-up | at month 2, 4, 6, 8, 10 and 12 after baseline
  A fall is defined as unintentional coming to rest on the ground, floor, or other lower level (coming to rest against furniture or a wall is not considered a fall). All reported incident falls will be ascertained every 2 month (phone calls at 2, 4, 8 and 10 months and clinical visits at 6 and 12 months after baseline) with a questionnaire evaluating the circumstances of each fall and injuries associated with it. Participants will also receive a diary to record any new health event including a fall. The diary will serve as a supplementary tool to falls evaluation minimizing potential recall bias.

SECONDARY OUTCOMES:
Number of participants who fell at least once during 12 months of follow up | at month 2, 4, 6, 8, 10 and 12 after baseline
Gait variability (stride time, stride length and gait speed) | Baseline, 6 & 12 months
  assessed by a GAITRite analysis system
Cognitive function | Baseline, 6 & 12 months
  assessed using the Montreal Cognitive Assessment (MoCA)
Alertness | Baseline, 6 & 12 months
  Alertness will be assessed using the two subtests "alertness" and "split alertness" of the test of attentional performance (TAP)
Quality of life | Baseline, 6 and 12 months
  evaluated using the SF-36 questionnaire

OTHER OUTCOMES:
progression of MCI/mild dementia | 6 &12 months
  any progression of the cognitive disorder to a more severe state ( will be confirmed based on medical records of the memory clinic of Waid City Hospital. Evaluation of this endpoint will be supported by information from the MoCA and the TAP subtests at baseline, 6, and 12 months clinical visits.
Musculoskeletal pain | baseline, 6 and 12 month
  assessed using McGill pain map. Number of painful joints will be assessed using a joint map.

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff-Ferrari, Prof., Principal Investigator — Director Geriatric Clinic University Hospital Zurich and Centre on Aging and Mobility, University of Zurich
Locations (1):
- Centre on Aging and Mobility, University of Zurich, Waid City Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Fischbacher M, Chocano-Bedoya PO, Meyer U, Bopp I, Mattle M, Kressig RW, Egli A, Bischoff-Ferrari HA. Safety and feasibility of a Dalcroze eurhythmics and a simple home exercise program among older adults with mild cognitive impairment (MCI) or mild dementia: the MOVE for your MIND pilot trial. Pilot Feasibility Stud. 2020 Jul 15;6:101. doi: 10.1186/s40814-020-00645-7. eCollection 2020. PMID 32695433